CLINICAL TRIAL: NCT04545853
Title: Associations Between Pain Perceptions and Movement-evoked Pain: a Cross-sectional Study.
Brief Title: Associations Between Pain Perceptions and Movement-evoked Pain.
Status: Withdrawn | Type: Observational
Why Stopped: Due to COVID-19
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Lynn Leemans, Principal Investigator, Vrije Universiteit Brussel
Other Study IDs: MEP_PC
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the associations between pain cognitions and movement-evoked pain in people with musculoskeletal pain complaints.

DETAILED DESCRIPTION:
This study will investigate the associations between pain cognitions and movement-evoked pain in people with musculoskeletal pain complaints. This study will be carried out as a cross-sectional study. Participants will be recruited by means of flyers and social media.

Pain cognitions will be assessed using questionnaires (The Pain Catastrophizing Scale (PCS), The llness perception questionnaire-revised (IPQ-R), The Pain Vigilance and Awareness Questionnaire (PVAQ), The Tampa Scale for Kinesiophobia (TSK), The 36-item short form health survey (SF-36)), whilst movement-evoked pain will be assessed using a lifting task. Participants will need to rate the experienced pain immediately after completing the task. To estimate the extent to which pain cognitions explain movement-evoked pain, correlational analyses will first be conducted between all variables to determine what variables will be included in the hierarchical regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* presence of musculoskeletal pain for more than three months,
* medically stable (no serious health conditions, no pending surgery or invasive medical procedure, no contraindication to physical activity).

Exclusion Criteria:

* Presence of co-existing pain conditions of other origins with chronic musculoskeletal pain not being the primary condition (i.e. predominant subject of symptom complaints)
* severe underlying comorbidity (like diagnosed diabetes, cardiovascular problems, etc.)
* pregnant or given birth in the preceding year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by flyers at the University Hospital Brussels, social media. Prior to inviting the eligible participants, the presence of musculoskeletal pain will be confirmed by phone in order to proceed to the informed consent process. Musculoskeletal pain is defined as pain, that potential participants report, feeling in the muscles, joints or bones. This pain can be localized, regional, or widespread.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Movement-evoked pain | Assessed only once at baseline.
  Pain that is experienced in response to a physical task. Participants will perform a lifting task. Participants will be asked to lift a series of 19-canisters that will be arranged in a standardized pattern on a waist-high table. Participants will provide a pain rating on a 11 points Numeric Rating Scale (NRS) with the endpoints no pain" (0) and "excruciating pain" (10)
Illness perceptions | Assessed only once at baseline
  The illness perception questionnaire-revised (IPQ-R) will be used to measure patients' illness perceptions. In the first domain, called illness identity, the perceived symptoms and their possible relation to the illness are evaluated. In this study, participants will indicate whether or not they believe that a specific symptom is related to pain ("yes" or "no"). The second domain, the beliefs domain, covers 7 dimensions: the acute/chronic timeline, the cyclical character of the illness, the consequences, controllability, curability, emotional representations and illness coherence. The third domain lists 18 possible causes to which individuals attribute their condition, the degree to which individuals perceive themselves as responsible for the illness, as well as the responsibility individuals take for curing themselves. For each item in the second and third domain, patients rate their level of agreement on a 5-point Likert scale, ranging from "strongly disagree" to "strongly agree"
Pain catastrophizing | Assessed only once at baseline
  The Pain Catastrophizing Scale (PCS) is a questionnaire to objectify catastrophic thinking about pain. It consists of 13 items describing different thoughts and feelings that individuals may have when experiencing pain. Items are scored on a 5-point scale. A general score and scores on 3 subscales (i.e., helplessness (6 items), magnification (3 items), and rumination (4items)) will be obtained; higher scores indicate more severe catastrophic thoughts about pain
Attention to pain | Assessed only once at baseline
  The Pain Vigilance and Awareness Questionnaire (PVAQ) will be used to investigate patients' attention to pain. It is a 16-item measure of attention to pain that assesses awareness, consciousness, vigilance, and observation of pain. Scores range from 0 to 80 and high scores correspond to hypervigilance for pain.
Fear of injury due to movement | Assessed only once at baseline
  The Tampa Scale for Kinesiophobia (TSK) is a 17-item questionnaire that will be used to measure the fear of (re) injury due to movement. Scores range from 17 to 68, with scores ≤ 37 suggesting low fear of movement and scores > 37 indicating high fear of movement.
Quality of life, an individual's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns. | Assessed only once at baseline
  The 36-item short form health survey (SF-36) is a multidimensional generic questionnaire assessing quality of life, which consists of 8 dimensions: physical functioning (10 items), role constraint caused by physical health problems (4 items), bodily pain (2 items), general health (5 items), vitality (4 items), social functioning (2 items), role constraint caused by emotional problems (3 items) and mental health (5 items). Higher scores reflecting a better health condition

IPD SHARING:
Plan to Share IPD: Undecided